CLINICAL TRIAL: NCT00337961
Title: Optic Nerve Sheath Fenestration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Karen Joos, Associate Professor of Ophthalmology, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 990379
Record Dates: First submitted 2006-06-16; First posted 2006-06-20 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Optic Nerve Sheath Fenestration
Keywords: Optic Nerve Sheath Fenestration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Optic Nerve Sheath Fenestration

SUMMARY:
The purpose of this study is to develop a way to perform safer surgery in the eye socket. The eye and its surrounding structures are very delicate and can easily be damaged from surgery. A laser may act as a gentle knife to cut the tissue. Currently, this is done with a small scissors and knife, but it could be done with gentle laser. By using an endoscope, the surgery could be much safer and faster. Vanderbilt has a Free Electron Laser, which could be used to make a small hole in the coverings around the optic nerve to treat certain diseases. Before it is used in seeing eyes, the laser must be tested on eyes which are to be removed during an enucleation to prove that it does not damage the optic nerve The standard enucleation (removal of your blind painful eye) will be performed. This procedure will be performed at the Free Electron Laser Center Operating Room, which is a fully equipped operating room currently being used for outpatient surgery. The post-operative recovery room setting is similar to the post-operative recovery room in the previously used area. This includes general anesthesia with a breathing tube in your throat, injecting an anesthetic liquid behind the eye for comfort after surgery, and removing the eyeball. Enucleations must be performed under general anesthesia or intravenous sedation with a retrobulbar injection (injection behind the eye). The anesthesiologist will determine which is safer to perform. The removed globe will be replaced with a spherical implant. Just prior to the removal of the eyeball, a small opening will be made in the coverings around your optic nerve (the cable exiting the eyeball) with the endoscopic laser or with a knife and scissors. The procedure should not take much longer than the standard eye removal. The procedure will be identical to the standard enucleation (eye removal) except for making the tiny hole in the coverings of the optic nerve, which should take about 15 to 30 minutes.

The laser is very tissue specific. It only reacts with certain types of tissue and should not damage the surrounding tissue.

There will be no additional costs to you associated with the study portion of the procedure.

DETAILED DESCRIPTION:
The purpose of this study is to develop a way to perform safer surgery in the eye socket. The eye and its surrounding structures are very delicate and can easily be damaged from surgery. A laser may act as a gentle knife to cut the tissue. Currently, this is done with a small scissors and knife, but it could be done with gentle laser. By using an endoscope, the surgery could be much safer and faster. Vanderbilt has a Free Electron Laser, which could be used to make a small hole in the coverings around the optic nerve to treat certain diseases. Before it is used in seeing eyes, the laser must be tested on eyes which are to be removed during an enucleation to prove that it does not damage the optic nerve The standard enucleation (removal of your blind painful eye) will be performed. This procedure will be performed at the Free Electron Laser Center Operating Room, which is a fully equipped operating room currently being used for outpatient surgery. The post-operative recovery room setting is similar to the post-operative recovery room in the previously used area. This includes general anesthesia with a breathing tube in your throat, injecting an anesthetic liquid behind the eye for comfort after surgery, and removing the eyeball. Enucleations must be performed under general anesthesia or intravenous sedation with a retrobulbar injection (injection behind the eye). The anesthesiologist will determine which is safer to perform. The removed globe will be replaced with a spherical implant. Just prior to the removal of the eyeball, a small opening will be made in the coverings around your optic nerve (the cable exiting the eyeball) with the endoscopic laser or with a knife and scissors. The procedure should not take much longer than the standard eye removal. The procedure will be identical to the standard enucleation (eye removal) except for making the tiny hole in the coverings of the optic nerve, which should take about 15 to 30 minutes.

The laser is very tissue specific. It only reacts with certain types of tissue and should not damage the surrounding tissue.

There will be no additional costs to you associated with the study portion of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Blind Eye Needing Enucleation

Exclusion Criteria:

* Capable of being performed at FEL Surgical OR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2000-07; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Histologic Evaluation | Measured at time of procedure
Ease of Procedure | At time of procedure
Histological Evaluation | At time of procedure

CONTACTS AND LOCATIONS:
Overall Officials: Sandy A Owings, COA, CCRP, Study Director — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States